CLINICAL TRIAL: NCT07296198
Title: Strongyloidiasis at CHRU Nancy: Evaluation of the Performance of Serological Tests and Disease-associated Characteristics
Acronym: SEROANGUILLULO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne DEBOURGOGNE, PU-PH, Central Hospital, Nancy, France
Other Study IDs: 2025PI080
Record Dates: First submitted 2025-11-26; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Strongyloidiasis
MeSH Terms: conditions — Strongyloidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Strongyloides serology — serological test for Strongyloides antibody

SUMMARY:
Strongyloidiasis is a disease caused by a parasite belonging to the helminth phylum: Strongyloides stercoralis. This nematode is mainly found in warm and humid regions, which favor its survival and transmission to humans. The disease presents several clinical forms: symptomatic forms, which are characteristic and make diagnosis easier, but also asymptomatic forms, where the parasite remains dormant in the human body thanks to the immune system. The latter form is particularly dangerous in cases of immunosuppression (cancers, corticosteroid treatment) or during organ donation. Therefore, knowing the serological status of a patient who has lived in an endemic area is essential to prevent severe strongyloidiasis.

To mitigate this risk, a new recommendation (2023) regarding the serological screening of organ donors has been issued, specifically concerning strongyloidiasis serology. To meet this requirement, the CHRU Nancy laboratory implemented an ELISA serological technique for detecting immunoglobulins directed against the parasite (Strongyloides stercoralis). A call for tenders was launched in summer 2025, with three responses from different suppliers (Launch, Euroimmun, Bordier).

Over the past 15 months, 600 serological tests have been performed, including 60 positive and 20 borderline results. The question is whether these results represent true strongyloidiasis cases and to assess the diagnostic performance of the technique used, particularly its specificity and sensitivity.

Primary objective:

Evaluate the performance of the three ELISA serological techniques for diagnosing strongyloidiasis.

Secondary objectives:

Identify and assess the socio-demographic, clinical, biological, and epidemiological characteristics of patients with strongyloidiasis.

Evaluate compliance with recommendations by healthcare professionals when faced with a positive strongyloidiasis serology (recommendations: add microfilaria serology and initiate ivermectin treatment).

Identify the context in which strongyloidiasis serology is prescribed (diagnosis of digestive parasitosis, compliance with PMO/organ recipient recommendations, pre-immunosuppression workup, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with strongyloidiasis serology performed between January 2024 and June 2025
* Whose serum tube residues are available in the biobank
* Who have not objected to the reuse of their data for research purposes

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with strongyloidiasis serology performed between January 2024 and June 2025
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
serological result | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France